EFFECT OF YOGA TRAINING ON CARDIOVASCULAR, AUTONOMIC, MENTAL HEALTH AND COGNITIVE PARAMETERS IN HYPERTENSIVE PATIENTS: A RANDOMIZED CONTROLLED CLINICAL TRIAL (Hypertension and Yoga – HY Study)

#### **ABSTRACT**

The objective of this study is to analyze the effect of 16 weeks of Yoga training on cardiovascular, autonomic, mental health, and cognitive parameters in hypertensive individuals. This is a randomized, controlled clinical trial conducted with adults and older adults (40 years or older), of both sexes, diagnosed with Arterial Hypertension (AH). They will be randomized into two groups: Yoga Group (YG) and Control Group (CG). The YG will undergo a 16-week Yoga training program involving breathing techniques, mobility, physical postures, relaxation, and meditation. In the first eight weeks (phase 1), three supervised sessions will be held weekly. In the last eight weeks of the study (phase 2), the training will consist of three supervised sessions per week and the delivery of an asynchronous video lesson, with the weekly frequency then increasing from three to four sessions per week. The video lesson will be available on a digital platform. Cardiovascular, autonomic, mental health, and cognitive parameters will be assessed before, after eight weeks, and after 16 weeks. Furthermore, the biomarkers brainderived neurotrophic factor (BDNF), serotonin, and nitric oxide will be analyzed at different study time points, as well as biochemical profile tests (glucose, total cholesterol, among others), functional capacity tests, and body composition. This project is expected to contribute to the literature by better elucidating the effects of yoga on the cardiovascular, mental, and cognitive health of hypertensive individuals. The SPSS (21.0) statistical package will be used for data analysis. After confirming the appropriate assumptions, generalized estimating equations will be used, followed by the Bonferroni post hoc test, with a significance level of 5%.

#### 1. INTRODUCTION

Systemic arterial hypertension (HA), characterized by high and sustained blood pressure (BP) levels, is a highly prevalent multifactorial disease in Brazil (BARROSO et al., 2021) and worldwide (FEITOSA et al., 2024). It is associated with the development of cardiovascular and cerebrovascular diseases, which currently lead the ranking of causes of mortality (LAVÔR et al., 2020). Furthermore, HA can impact mental health and brain structure and function, leading to a greater likelihood of developing depressive and anxious symptoms and impaired cognitive functions, with impairment of executive functions, inhibitory control, attention, and memory, and a greater risk of developing dementia (RÊGO et al., 2019). In this sense, it is emphasized that the treatment of HA should focus not only on improving aspects of the patient's cardiovascular health, but also their mental and cognitive health. In addition to pharmacological treatment, lifestyle changes are recommended, with emphasis on regular physical exercise. Several organizations, such as the American College of Sports Medicine, the Brazilian Society of Hypertension, and the European Society of Cardiology (WHELTON ET AL., 2017; BARROSO et al., 2021; CAREY et al., 2022), unanimously recognize the role of physical training, particularly aerobic and resistance training, in the management of hypertension. Indeed, the literature consistently demonstrates the benefits of these two types of physical training in reducing chronic BP (MACDONALD; PESCATELLO, 2018; WHELTON ET AL., 2017; EDWARDS ET AL., 2023).

However, many hypertensive individuals do not adhere to the recommended conventional physical training programs. In Brazil, data indicate that only 26.9% of patients with hypertension perform at least 150 minutes of moderate physical activity or 75 minutes of vigorous activity per week (SZWARCWALD et al., 2021). Therefore, it is necessary to focus on unconventional forms of physical exercise, as these can often be more attractive. In this scenario, Yoga presents itself as an alternative, as it has been gaining more followers and has been identified as an attractive practice, especially among those who have barriers to adherence to conventional physical training (BRINSLEY et al., 2019). The literature has indicated that Yoga, through breathing control, relaxation, and meditation techniques, can help reduce mental stress, improve well-being, and improve symptoms of anxiety and depression (A'NAJA et al., 2024; BRINSLEY et al., 2021). Furthermore, studies indicate the potential of Yoga to promote improvements in cardiovascular parameters, such as lowering blood pressure and improving

vascular function (AHUJA et al., 2024; PATIL et al., 2024). Furthermore, it is a safe, low-cost practice widely practiced worldwide, especially in the West (THOMAS et al., 2021; BRINSLEY et al., 2019).

However, there is a clear lack of more robust studies investigating the effects of Yoga on cardiovascular, autonomic, mental health, and cognitive parameters, especially in hypertensive individuals. Furthermore, it is necessary to investigate the mechanisms that explain the possible reduction in blood pressure and the improvement in mental and cognitive health of hypertensive individuals resulting from Yoga training.

The development of this study is expected to better understand the effects of Yoga training, as a potential unconventional modality, on cardiovascular, autonomic, mental health, and cognitive parameters in adults and older adults with hypertension. If its positive effects are proven, yoga could be considered an interesting alternative physical exercise practice to complement comprehensive hypertension treatment.

Thus, the following research question arose: what are the effects of 16 weeks of yoga training on cardiovascular, autonomic, mental health, and cognitive parameters in hypertensive individuals

#### 1.1 OBJECTIVES

## 1.1.1 General Objective

To analyze the effect of 16 weeks of Yoga training on cardiovascular, autonomic, mental health and cognitive parameters in hypertensive patients.

### 1.1.2 Specifics objectives

- Analyze the effect of eight and 16 weeks of Yoga training on clinical and ambulatory blood pressure, vascular function, heart rate variability, and cerebral blood flow in hypertensive individuals.
- Analyze the effect of eight and 16 weeks of Yoga training on depressive symptoms, anxiety, stress, sleep quality, and quality of life in hypertensive individuals.
- Analyze the effect of eight and 16 weeks of Yoga training on cognitive function and attention span in hypertensive individuals.

- Analyze the effect of eight and 16 weeks of Yoga training on serum levels of BDNF, cortisol, and nitric oxide in hypertensive individuals.
- Analyze the effects of eight and 16 weeks of Yoga training on the biochemical profile (glucose, total cholesterol, HDL cholesterol, triglycerides, aspartate aminotransferase, alanine aminotransferase, and creatinine) in hypertensive individuals.
- Analyze the effects of eight and 16 weeks of Yoga training on functional capacity (flexibility and strength) in hypertensive individuals.
- Analyze the effects of eight and 16 weeks of Yoga training on body composition in hypertensive individuals.
- Correlate the potential changes identified in blood pressure resulting from Yoga training with the potential changes observed in heart rate variability, vascular function, and serum nitric oxide concentrations in hypertensive individuals.
- Correlate the potential changes identified in mental health resulting from Yoga training with the potential changes observed in cardiovascular parameters and serum cortisol concentrations in hypertensive individuals.
- Correlate the potential changes identified in cognitive function resulting from Yoga training with the potential changes observed in cardiovascular parameters and BDNF in hypertensive individuals.
- Develop a digital platform that allows access to online Yoga classes (second phase of the intervention) via a mobile app and/or website.

#### 2 METHODS

#### 2.1 STUDY DESIGN

This is a randomized and controlled clinical trial to be conducted in parallel at the Sports Center (CDS), at the Federal University of Santa Catarina (UFSC) (Florianópolis) and which will be registered in Clinical Trials and the Brazilian Clinical Trials Registry (Rebec).

#### 2.2 PARTICIPANTS

Seventy adults or elderly individuals (>= 40 years), of both sexes, diagnosed with hypertension controlled by up to three medications, who do not present high cardiovascular risk (RIEBE et al., 2015) and have not engaged in a physical exercise program in the six months prior to the start of the study will participate in the study. The exclusion criteria will be: adherence to less than 75% of training sessions; diagnosis of other diseases during the study; adherence to another physical exercise program; change in the class and/or dose of antihypertensive medication during the study; worsening of the disease (resting systolic blood pressure (BP) > 180 mmHg). Recruitment will be based on advertising in local media and posting of posters in the vicinity of public hospitals.

### 2.3 ETHICAL ASPECTS

This study is guided by Resolution 466/2012 and will be submitted to the UFSC Human Research Ethics Committee. All interested volunteers will participate in an initial meeting where the project will be explained, including all procedures, the risks and benefits of participating in this study, and information that they may withdraw from the study at any time. Volunteers who meet the eligibility criteria will be invited to read and, if they agree, sign the Informed Consent Form (ICF) to participate in this study.

#### 2.4 ALOCATION AND RANDOMIZATION

Participants will be randomly assigned to two groups: Yoga Group (YG) and Control Group (CG). Randomization will be performed 1:1 based on sex and mean systolic BP through

the website www.randomizer.org by an independent researcher not involved in the assessments or intervention. The allocation list will be hidden from all evaluators until the end of the study.

#### 2.4 EXPERIMENTALS PROCEDURE

Before, during, and after the study, participants will undergo assessments. For this research, data collected during anamnesis (APPENDIX A) will be analyzed to characterize the sample. Additionally, cardiovascular and autonomic assessments will be performed, as well as mental health, cognitive function and attention, biochemical markers, functional capacity, body composition, and control variables such as anthropometry. Specifically for the GY, indicators of internal training load, affective response, and acute blood pressure responses will be collected in some training sessions.

#### 2.5 OUTCOMES

## 2.5.1 Sample characteristics

For the purpose of characterizing the sample, sociodemographic data (sex and age), health condition data (diseases, time of diagnosis, type, frequency and dosage of medications used) and lifestyle data (smoking, alcohol use, level of habitual physical activity, time of engagement in the program) will be collected from an anamnesis.

### 2.5.2 Cardiovascular and autonomic parameters

Clinical BP will be measured using an Omron HEM 742 oscillometric device (OMRON Healthcare, Kyoto, Japan), according to current recommendations. Ambulatory BP will be assessed over 24 hours using a Dyna-MAPA device (Cardios), both in accordance with current recommendations (FEITOSA et al., 2024).

Vascular function will be assessed using the flow-mediated dilation technique following the recommendations of Thijssen et al. (2019), and cerebral blood flow will be estimated by measuring blood flow in the internal carotid artery (THOMAS et al., 2015), both using a LOGIQ S7 Expert Ultrasound (GE Healthcare). Data analysis will be performed using FMD Studio software (Cardiovascular Suite, Quipu version 4.2.1, Italy). Cardiac autonomic

modulation will be assessed by heart rate variability, following current recommendations (TASK FORCE, 1996). After collection, the RR intervals will be exported to the Kubios HRV program (Biosignal Analysis and Medical Imaging Group, Finland), whose analyses will be performed in the time and frequency domains (TASK FORCE, 1996).

### 2.5.3 Mental health parameters

Quality of life will be assessed using the EQ-5D-5L (ANNEX A) and Short Form-36 (ANNEX B) questionnaires. The EQ-5D-5L consists of five domains, with lower scores indicating better quality of life. It also contains a health perception scale, where 0 represents the worst health and 100 represents the best health (EUROQOL, 2025). The SF-36 is multidimensional and consists of 36 items, grouped into eight domains. It has a score ranging from 0 to 100 (VAN ROTTERDAM, HENSLEY, HAZELTON, 2021).

Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI-BR) (ANNEX C), a 19-question questionnaire. The questions are grouped into seven components, with scores above 5 indicating poor sleep quality (BERTOLAZI et al., 2011; BUYSSE, 1989).

Depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9) (ANNEX D), consisting of nine questions, yielding an overall score ranging from 0 to 27 points (APA, 2000; SANTOS et al., 2013), and the Hospital Anxiety and Depression Scale (HAD) (ANNEX E), consisting of 14 multiple-choice items, with an overall score ranging from 0 to 21 (BOTEGA et al., 1995).

Perceived stress will be assessed using the Perceived Stress Scale-10 (PSS-10) (ANNEX F), intended to provide a global measure of stress. Scores range from 0 to 40 points. Higher scores represent a higher level of perceived stress (SIQUEIRA REIS, FERREIRA HINO & RODRIGUEZ AÑEZ, 2010).

## 2.5.4 Cognitive function and attention parameters

Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA) questionnaire (ANNEX G), which comprises eight domains. The maximum score is 30 points, corresponding to the best cognitive ability (HOBSON, 2015).

The Stroop Test (ANNEX H) will assess attention and inhibitory response capacity, calculating response time and accuracy. Better results are associated with shorter response times and fewer errors. By comparing congruent and incongruent conditions, cognitive interference and inhibitory control will be assessed (STROOP, 1935).

### 2.5.5 Biochemical markers parameters

Venous blood samples will be collected during fasting for analysis of cognitive and cardiovascular health biomarkers—BDNF, cortisol, and nitric oxide—at the Clinical Biochemistry Research Laboratory (CCS/UFSC). Serum cortisol and BDNF levels will be determined using enzyme-linked immunosorbent assays (ELISA) according to the manufacturer's instructions (BD Biosciences Pharmingen, San Diego, CA), with a detection limit of 2.2 pg/mL. Plasma nitric oxide concentrations will be measured using chemiluminescence, which allows for the accurate quantification of nitric oxide levels through conversion to nitrates and nitrites.

In addition, biochemical profile markers will be analyzed: glucose, total cholesterol, HDL cholesterol, triglycerides, aspartate aminotransferase, alanine aminotransferase, and creatinine. From the serum, all these markers will be dosed, using the respective method, in the BS 120 automation equipment, Mindray® using the available reagent kit, following the manufacturer's instructions.

## 2.5.6 Functional capacity parameters

Strength and flexibility tests will be performed to assess functional capacity.

The strength tests will be Handgrip Strength (HGS) and Isometric Muscle Strength of the Upper and Lower Limbs.

Isometric HGS will be measured using a Carci @— hydraulic dynamometer (CEFISE, São Paulo, SP). The patient will be seated with the arm in shoulder adduction, elbow flexed at 90°, and forearm in a neutral position. The participant will be asked to exert the greatest possible force by squeezing the dynamometer for five seconds. Three measurements will be taken on both sides, with a one-minute interval between each, and the highest value recorded in kilograms-force (kgf).

The maximum isometric force production capacity of the elbow and knee flexor and extensor muscle groups will be assessed using a microFET2 HHD digital dynamometer (Hoggan Health Industries, Salt Lake City, Utah). For upper limb measurements, the participant will be positioned on a stretcher in the supine position, with the shoulder joint adducted, the elbow flexed at 90°, and the forearm in a neutral position. For the lower limbs, the participant will be seated on the stretcher, with the knees flexed at 90°. Once positioned, the participant

will be instructed to exert force against the evaluator, who will hold the dynamometer for five seconds.

This process will be repeated three times on each side, for both the lower and upper limbs, with a 30-second interval between each contraction. The result will be recorded in kilograms-force (kgf). The 90° position angle of the elbow and knee joints will be determined using a universal goniometer with two 20 cm long rods and a fulcrum with a measurement accuracy of two degrees (Trident Gon-PVC).

To measure flexibility, the Sit and Reach Test, from the Senior Fitness Test battery (RIKLI; JONES, 2013), will be used, using the Wells bench. The participant will sit on a mat with both knees extended and their heels touching the bench. Without bending their knees, they will place one hand on top of the other and flex their hips so that the torso projects forward and the participant can push the ruler marked on the bench as far as it will go. Each participant will be given two attempts, and the highest score will be considered.

### 2.5.7 Body composition parameters

Using dual-energy X-ray absorptiometry (DXA), a Lunar Prodigy Advance (General Electric-GE®, Diegem, Belgium), fat mass, fat-free mass, lean mass, and bone mineral density will be assessed, all as a function of total density and expressed in absolute and relative terms. The device will be calibrated and used according to the manufacturer's recommendations.

Phase angle (PhA) will be estimated using bioimpedance, a multifrequency InBody® 720 (Biospace, Los Angeles, USA), with eight electrodes, measuring resistance at five frequencies (1, 50, 250, 500, and 1000 kHz) and reactance at three (5, 50, and 250 kHz). To estimate PhA, the raw BIA values will be used: resistance (R) and reactance (Xc). The technique provides impedance (Z) and Xc data at a frequency of 50 kHz, and from these, the R value will be calculated by the proportional sum of the body, in which the upper limbs represent 40% of the total body R, the trunk represents 10% and the lower limbs represent 50%. Thus, the PhA, expressed in degrees (O), will be calculated through the equation: PhA = Arctangent (Xc / R) \* (180 /  $\pi$ ) (NORMAN et al., 2012). The device will be calibrated and used according to the manufacturer's recommendations.

#### 2.5.8 Control outcomes

The following control variables will be collected: a) anthropometry (height, body mass, waist circumference), b) adherence to medication treatment (Morisky Therapeutic Adherence Scale) (ANNEX I) (OLIVEIRA-FILHO et al., 2012); c) habitual physical activity (accelerometry) and d) eating habits (Food Frequency Questionnaire) (ANNEX J).

#### 2.6 INTERVENTION

The intervention will last 16 weeks, with assessments before, after eight weeks, and after 16 weeks of cardiovascular, autonomic, mental health, and cognitive parameters, as well as control variables.

The YG will receive an intervention involving Yoga Training (YT), which will be divided into two phases: Phase 1 (first eight weeks), which will be supervised, with three weekly sessions lasting 60 minutes; and Phase 2 (the following eight weeks), which will consist of three supervised sessions per week and an asynchronous video lesson delivered via a digital platform, with an increment of one session per week. The classes will also be 60 minutes long. The supervised sessions will take place at the UFSC CDS rehabilitation center.

The YT sessions will follow the following structure: breathing techniques (Pranayama), warm-up (Pavana Muktasana), physical postures in standing, sitting, and lying positions (Asanas), and relaxation (Yoganidrá). The postures will be prescribed by holding time in seconds (30 to 40 seconds), number of sets, and rest between sets. Each session will include beginner, intermediate, and advanced postures. Furthermore, to reduce training monotony and contribute to affective and adherence to TY, elements of the breathing techniques and relaxation sections will be modified each session, and the postures will be modified each week. TY will progress throughout the intervention period, as follows:

- 1st progression (from the first four weeks to the second four weeks) □ increase in the number of physical postures in the standing position, considering that, in this group of postures, strength and balance predominate. Therefore, remaining in these postures for longer periods results in progression, with an increase in session intensity. To maintain the total session time, the warm-up and lying-down postures will be reduced.
- 2nd progression (from the first eight fully supervised weeks to the second eight weeks with the addition of video classes) □ progression in weekly frequency, from three sessions per

week to four sessions per week, with one of these sessions being via asynchronous video classes. Participants can choose the best day and time for the class, based on their routine.

- 3rd progression (transition to the last four weeks of intervention) □ further increase in the volume of standing postures, even greater than in the first progression. To maintain the total session time, the volume of warm-up and lying postures will be reduced.

The CG will not receive any intervention during the study and, like the SG participants, will be instructed not to change their routines. After the study period, the CG will be invited to participate, free of charge, in an exercise program similar to the one offered to the SG or another exercise program aimed at this population that is already offered at the Sports Center. Additionally, the GC will also have access to video lessons through the digital platform.

It is important to note that the project activities will be led by properly trained graduate students in Physical Education, with the assistance of undergraduate Physical Education students, under the supervision of the professors involved in the project.

#### 2.7 MONITORING AND SAFE

During the GY training sessions, safety, load, and affectivity monitoring information will be collected. For safety purposes, blood pressure will be measured before the start of each session, respecting the cutoff values for physical exercise: values greater than 160 mmHg for systolic blood pressure and/or 105 mmHg for diastolic blood pressure.

The internal workload of each training session will be quantified by the Subjective Perceived Exertion (RPE) (ANNEX K) of the session, using the scale adapted from Borg (FOSTER et al., 2001), aiming to estimate the intensity after each exercise session, with individual questions after the sessions. Exercise affectivity will be assessed using the Hardy and Rejeski sensation scale (HARDY and REJESKI, 1989) (ANNEX L), with 11 points ranging from +5 (very good) to -5 (very bad), with patients answering the following question at the end of the session: "How pleasant was it for you to carry out this exercise session?".

#### 2.8 ADVERSES EVENTS

Participants will be monitored throughout the study for adverse events using a standardized form. For GY participants, this information will be collected weekly, while for CG participants, this form will be completed midway through and at the end of the study period. The possibility of discontinuation from the study will be discussed by the study coordinators

and management in the event of a serious adverse event or a series of mild to moderate adverse events.

### 2.9 DATA ANALYSIS

Data will be analyzed using SPSS (21.0), adopting a 5% significance level. The general characteristics of the study participants will be presented with measures of central tendency and dispersion (numerical variables), or absolute and relative frequency (categorical variables), depending on the data distribution, to be verified using the Shapiro-Wilk test. After confirming the appropriate assumptions, Generalized Estimating Equations will be used, followed by the Bonferroni post-hoc test, to identify possible intra- and intergroup differences throughout the study.

#### REFERENCES

AHUJA, Navdeep et al. Yoga Nidra for hypertension: A systematic review and meta-analysis. Journal of Ayurveda and Integrative Medicine, v. 15, n. 2, p. 100882, 2024.

AMERICAN PSYCHIATRIC ASSOCIATION et al. Diagnostic and statistical manual of mental disorders. Text revision, 2000.

A'NAJA, M. Newsome et al. 2024 ACSM Worldwide Fitness Trends: Future Directions of the Health and Fitness Industry. ACSM's Health & Fitness Journal, v. 28, n. 1, p. 14-26, 2024.

BARROSO, Weimar Kunz Sebba et al. Diretrizes brasileiras de hipertensão arterial–2020. Arquivos brasileiros de cardiologia, v. 116, p. 516-658, 2021.

BERTOLAZI, A. N. et al. Validation of the Brazilian Portuguese version of the Pittsburgh sleep quality index. Sleep medicine, v. 12, n. 1, p. 70-75, 2011.

BOTEGA, N. J. et al. Mood disorders among inpatients in ambulatory and validation of the anxiety and depression scale HAD. Revista De Saúde Pública, v. 29, n. 5, p. 355–363, 1995.

BRINSLEY, Jacinta et al. Effects of yoga on depressive symptoms in people with mental disorders: a systematic review and meta-analysis. British journal of sports medicine, v. 55, n. 17, p. 992-1000, 2021.

BUYSSE, Daniel J. et al. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry research, v. 28, n. 2, p. 193-213, 1989.

CAREY, Robert M.; MORAN, Andrew E.; WHELTON, Paul K. Treatment of hypertension: a review. Jama, v. 328, n. 18, p. 1849-1861, 2022.

EDWARDS, Jamie J. et al. Exercise training and resting blood pressure: a large-scale pairwise and network meta-analysis of randomised controlled trials. British Journal of Sports Medicine, v. 57, n. 20, p. 1317-1326, 2023.

ELECTROPHYSIOLOGY, Task Force of the European Society of Cardiology the North American Society of Pacing. Heart rate variability: standards of measurement, physiological interpretation, and clinical use. Circulation, v. 93, n. 5, p. 1043-1065, 1996.

EUROQOL. *EQ-5D-5L*. Disponível em: <a href="https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-5l/">https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-5l/</a>. Acesso em: 10 de abril de 2025.

FEITOSA, Audes Diogenes de Magalhães et al. Diretrizes Brasileiras de Medidas da Pressão Arterial Dentro e Fora do Consultório–2023. Arquivos Brasileiros de Cardiologia, v. 121, p. e20240113, 2024.

FOSTER, C. et al. A new approach to monitoring exercise training. Journal of Strength and Conditioning Research, v. 15, n. 1, p. 109-115, 2001.

HARDY CJ, REJESKY WJ. Not what, but how one feels: the measurement of afect during exercise. J Sport Exerc Psychol. 1989;11:304–17.

HOBSON, John. The montreal cognitive assessment (MoCA). Occupational Medicine, v. 65, n. 9, p. 764-765, 2015.

LAVÔR, Layanne Cristina de Carvalho et al. Prevalence of arterial hypertension and associated factors: a population-based study. Revista da Associação Médica Brasileira, v. 66, p. 630-636, 2020.

MACDONALD, Hayley V.; PESCATELLO, Linda S. Exercise prescription for hypertension: new advances for optimizing blood pressure benefits. In: Lifestyle in heart health and disease. Academic Press, 2018. p. 115-136.

OLIVEIRA-FILHO, Alfredo Dias et al. Relação entre a Escala de Adesão Terapêutica de oito itens de Morisky (MMAS-8) e o controle da pressão arterial. Arquivos Brasileiros de Cardiologia, v. 99, p. 649-658, 2012.

PATIL, Satish G. et al. Effect of yoga on endothelial function: A systematic review and metaanalysis. Journal of Integrative and Complementary Medicine, v. 30, n. 3, p. 233-249, 2024.

RÊGO, Maria LM et al. Physical exercise for individuals with hypertension: it is time to emphasize its benefits on the brain and cognition. Clinical Medicine Insights: Cardiology, v. 13, p. 1179546819839411, 2019.

RIEBE, Deborah et al. Updating ACSM's recommendations for exercise preparticipation health screening. 2015.

RIKLI, RE.; JONES, C.J. Senior fitness test manual. California: Human Kinetics, 2013.

SANTOS, Iná S. et al. Sensibilidade e especificidade do Patient Health Questionnaire-9 (PHQ-9) entre adultos da população geral. Cadernos de saúde pública, v. 29, p. 1533-1543, 2013.

SIQUEIRA REIS, Rodrigo; FERREIRA HINO, Adriano Akira; ROMÉLIO RODRIGUEZ AÑEZ, Ciro. Perceived stress scale: Reliability and validity study in Brazil. Journal of health psychology, v. 15, n. 1, p. 107-114, 2010.

STROOP, J. Ridley. Studies of interference in serial verbal reactions. Journal of experimental psychology: General, v. 18, p. 643-662, 1935.

SZWARCWALD, Célia Landmann et al. Healthy lifestyle and recommendations in health care among hypertensive and diabetic patients in Brazil, 2019. Revista Brasileira de Epidemiologia, v. 24, p. e210017, 2021.

THIJSSEN, Dick HJ et al. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. European heart journal, v. 40, n. 30, p. 2534-2547, 2019.

THOMAS, Allie et al. The integration of yoga in physical therapy clinical practice. Complementary therapies in medicine, v. 59, p. 102712, 2021.

THOMAS, Kate N. et al. Technical recommendations for the use of carotid duplex ultrasound for the assessment of extracranial blood flow. American Journal of Physiology-Regulatory, Integrative and Comparative Physiology, v. 309, n. 7, p. R707-R720, 2015.

VAN ROTTERDAM, Flora-Joan; HENSLEY, Michael; HAZELTON, Michael. Measuring change in health status over time (responsiveness): a meta-analysis of the SF-36 in cardiac and pulmonary rehabilitation. Archives of rehabilitation research and clinical translation, v. 3, n. 2, p. 100127, 2021.

WHELTON, Paul K. et al. Acc/aha/aapa/abc/acpm/ags/APhA/ASH/ASPC/nma/pcna guideline for the prevention, Detection, evaluation, and management of high blood pressure in adults: a Report of the American College of Cardiology/American heart Association. Task force on clinical practice guidelines//J. Am. Coll. Cardiol.-2017.-Nov 13. Почки, v. 7, n. 1, p. 68-74, 2018.

## APPENDIX

## **APPENDIX A** – Anamnesis

| I) DADOS SOCIODEMOGRÁFICOS | |
|---|---|
| 1) Nome completo: | |
| 2) Endereço: | |
| 3) Telefone de contato: Celular: | |
| 4) Data de nascimento: | |
| 5) Estado civil: ( ) casado (a)/união consensual ( ) solteiro (a) | |
| ( )Separado (a)/ divorciado (a)/ desquitado (a) ( )viúvo (a) | |
| 6) Grau de escolaridade: ( ) fundamental incompleto ( ) fundamental completo | |
| ( )ensino médio incompleto ( ) ensino médio completo ( ) superior incompleto ( ) super | ioi |
| 7) Qual é a sua principal ocupação (Ocupação que gera maior renda): | |
| II) HISTÓRICO DE SAÚDE | |
| II.1) Algum médico já lhe disse que você tem ou já teve: ( Entrevistador, leia as opções). | |
| II.1.1) Doença arterial coronariana (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.2) Hipertensão arterial/ pressão alta (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.3) Diabetes (açúcar no sangue) (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.4) Colesterol e/ou Triglicérides alto (gordura no sangue) (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.5) Doença pulmonar (asma, enfisema, DPOC, etc) (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.6) Coração grande ou já fez transplante cardíaco (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.7) Arritmias, disritmias, falha no coração (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.8) Aneurisma, derrame ou acidente vascular cerebral (0) Não (1) Sim Há quanto | |
| tempo? | |
| II.1.9)Problema nas válvulas do coração (0) Não (1) Sim Há quanto | |
| tempo? | |

| II.1.10)Doença de Chagas (0) Não (1) Sim Há quanto |
|---|
| tempo? |
| Outras doenças ou problemas de saúde? Está sob acompanhamento médico? (0) Não (1) Sim Sente dores no peito (angina)?Se sim, com que cia? al(is) medicamento(s) você utiliza regularmente (Informar nome, indicação, dose, cia semanal e horário do dia)? Há alguma queixa ou dúvida em relação aos nentos em uso? cê possui alguma limitação física (dor, lesão ou cirurgia nos ossos, músculos ou ções) que limite e/ou impeça a prática de atividades físicas? |
| quanto tempo? |
| II.1.12) Outras doenças ou problemas de saúde? |
| II.1.13) Está sob acompanhamento médico? (0) Não (1) Sim II.2) Sente dores no peito (angina)?Se sim, com que frequência? |
| II.3) Qual(is) medicamento(s) você utiliza regularmente (Informar nome, indicação, dose frequência semanal e horário do dia)? Há alguma queixa ou dúvida em relação ao medicamentos em uso? |
| II.4) Você possui alguma limitação física (dor, lesão ou cirurgia nos ossos, músculos o articulações) que limite e/ou impeça a prática de atividades físicas? |
| II 5) Duranto a prática do atividado física você já sontiu algum dossos sintomas? |
| 1.Dor ou desconforto no peito (0) Não (1) Sim |
| 2.Falta de ar durante exercício leve (0) Não (1) Sim |
| 3.Tontura ou desmaio (0) Não (1) Sim |
| 4.Palpitação ou taquicardia (0) Não (1) Sim |
| 5.Dor nas pernas quando caminha (0) Não (1) Sim |
| 6.Cansaço grande para atividadesleves (0) Não (1) Sim |
| (1) S.M. |
| II.6)Algum parente (primeiro grau) já teve problema cardíaco? (0) Não (1) Sim (7) Não Sabe |
| II.7)Atualmente, você fuma cigarros? (0) Não (1) Sim |

| II.7.1) Se sim, em mé | dia quantos cigarros você fuma por dia? cigarros (7) Não sabe |
|---|---|
| (8) NA | |
| III) PRÁTICA DE E | XERCÍCIOS FÍSICOS |
| III.1) Atualmente, vo | cê pratica alguma atividade física de maneira regular (pelo menos |
| 2 vezes por semana)? | não sim |
| III.1.1) Se sim, por fa | vor, especifique: |
| corrida | hidroginástica caminhada |
| futebol | musculação ginástica |
| natação | outro (especifique) |
| III.1.2) Total de min | utos dispendidos em atividades nestas atividades elencadas acima, |
| por semana: | |
| 40-60 minutos | /semana |
| 61-80 minutos | /semana |
| 81-100 minuto | os/semana |
| 100 ou mais n | inutos/semana |

## APPENDIX B

## FICHA DE CONTROLE SEMANAL – SINTOMAS E/OU EVENTOS ADVERSOS

| ID participante/nome: | Data: |
|---|---|
| Semana de treino | |
| Profissional: | |
| MUDANÇA DE HÁBITOS NOS ÚL | ΓΙΜΟS 7 DIAS. |
| Realizou alguma atividade física fora | do habitual? ( ) Sim ( ) não |
| | L-ESTAR DURANTE OU APÓS AS SESSÕES DE |
| TREINAMENTO NOS ÚLTIMOS 7 | |
| Desconforto respiratório ( ) Sim ( ) | ) não |
| Associado ao exercício ( ) Sim ( ) | |
| Se sim: ( ) Durante as sessões ( ) L | ogo após as sessões ( ) Em domicílio |
| Desconforto muscular ( ) Sim ( ) | não |
| Dor muscular tardia ( ) | |
| Associado ao exercício ( ) Sim ( ) | não |
| Se sim: ( ) Durante as sessões ( ) L | ogo após as sessões ( ) Em domicílio |
| Desconforto articular Sim ( ) não | ( ) |
| Associado ao exercício Sim ( ) não ( | |
| Se sim: ( ) Durante as sessões ( ) L | ogo após as sessões ( ) Em domicílio |
| Outros ( ) | |

| DURANTE OU APÓS AS SESSÕES DE |
|------------------------------------|
| ( ) não |
| ( ) Náusea e/ou vômito |
| ( ) Palpitação |
| ( ) Visão turva/embaçada |
| ( ) Falta de ar |
| perglicêmica ( ) Crise hipotensiva |
| iva ( ) Crise respiratória |

| Associado ao exercício? ( ) Sim ( ) não | - |
|------------------------------------------------------|---|
| Necessitou de internação hospitalar? ( ) Sim ( ) não | |

#### APPENDIX C



#### TERMO DE CONSENTIMENTO LIVRE E ESCLARECIDO

Título: EFEITO DO TREINAMENTO DE YOGA SOBRE PARÂMETROS
CARDIOVASCULARES, AUTONÔMICOS, DE SAÚDE MENTAL E COGNITIVA EM
HIPERTENSOS: UM ENSAIO CLÍNICO RANDOMIZADO E CONTROLADO
(Hypertension and Yoga – HY Study)

**Pesquisador responsável:** Prof<sup>a</sup>. Dr<sup>a</sup>. Aline Mendes Gerage da Silva (CDS/ UFSC)

Você está sendo convidado a participar deste estudo que está vinculado a um projeto de tese do Programa de Pós-Graduação em Educação Física da Universidade Federal de Santa Catarina. Se você decidir fazer parte do estudo, precisará saber das possibilidades de riscos e benefícios e confirmar sua participação por meio deste termo de consentimento livre e esclarecido. Este documento esclarece sobre o estudo que você deseja participar. Se você tiver qualquer pergunta, por favor, sinta-se à vontade para entrar em contato com a equipe responsável pela condução do estudo que vamos esclarecer suas dúvidas. Esta pesquisa está pautada na Resolução 466/2012, do Conselho Nacional de Saúde e os pesquisadores comprometem-se em cumprir todos os seus itens.

A decisão de fazer parte do estudo é **voluntária** e você pode recusar ou retirar-se do estudo a qualquer momento sem nenhum tipo de prejuízo.

O **objetivo** dessa pesquisa é analisar o efeito de 16 semanas do treinamento de Yoga sobre parâmetros cardiovasculares, autonômicos, de saúde mental e cognitiva em hipertensos.

Justificativa: A pesquisa se justifica pela necessidade de preencher uma lacuna significativa na literatura científica sobre como uma modalidade não convencional como a Yoga pode atuar diante dos aspectos dessa doença crônica não transmissível altamente prevalente, considerando os componentes da modalidade Yoga (técnicas respiratórias, posturas físicas e relaxamento), fornecendo dados concretos que podem subsidiar a implementação de políticas de saúde direcionadas. Além disso, busca-se contribuir para a melhoria da qualidade de vida e bem-estar das pessoas com Hipertensão Arterial.

Procedimentos da Fase Experimental: Os procedimentos da pesquisa ocorrerão conforme especificado a seguir.

- Após se voluntariar para o estudo o(a) senhor(a) passará por uma entrevista inicial, com uma triagem a fim de identificar se você se encaixa no perfil do nosso estudo. Caso seja selecionado, o(a) senhor(a) será convidado a preencher e assinar o presente termo de consentimento, bem como a ficha de anamnese.
- Após a finalização da primeira etapa, o(a) senhor(a) será direcionado(a) para o agendamento das avaliações antecedentes ao início do projeto, a citar: a) medidas da pressão arterial, dos batimentos do coração e avaliação da saúde das suas artérias; b) questionários que avaliam seu estilo de vida, sua qualidade de vida, sua qualidade do sono e alguns sentimentos e capacidade cognitiva e memória; c) exames de sangue que avaliam o seu perfil metabólico e inflamatório; d) medidas de peso, estatura, composição corporal e outros parâmetros de medidas corporais; e) medidas de capacidade funcional (flexibilidade e força) e f) avaliação do nível de atividade física por um aparelho portátil a ser colocado em sua cintura. Essas avaliações acontecerão durante uma semana, em dias alternados e, em cada dia, o (a) senhor (a) gastará no máximo 2 horas. Depois de oito e 16 semanas do estudo, as avaliações iniciais serão repetidas, em semanas destinadas exclusivamente a essas avaliações.
- -Após as avaliações iniciais, haverá um sorteio para definir qual grupo você fará parte. Se você for sorteado para o grupo intervenção, você participará de um programa de treinamento físico, que envolverá a realização da modalidade Yoga em três a quatro vezes por semana. Caso você seja sorteado para o grupo controle, ao término do estudo, será convidado a participar de maneira gratuita de um programa de exercícios semelhante ao oferecido ao grupo intervenção ou outro programa de exercícios oferecido no Centro de Desportos. Também ao término do estudo, todos os participantes receberão o relatório completo de todas as avalições às quais forem submetidos e as vídeo-aulas de Yoga.

Desconforto ou Riscos Esperados: As coletas serão realizadas por pesquisadores da área da saúde, experientes e capacitados para cada medida. Entretanto, alguns desconfortos podem ocorrer. De maneira geral, pode-se esperar: um ligeiro incômodo no braço durante as medidas de pressão arterial, função vascular e durante a coleta de sangue. Especificamente para avaliações que deverão ocorrer em estado de jejum, os pesquisadores disponibilizarão um lanche logo após o término da coleta com objetivo de minimizar desconforto associado ao jejum. Este lanche será de responsabilidade e custeio dos pesquisadores. Se por ventura você apresentar algum sintoma/desconforto anormal durante alguma avaliação ou no decorrer da

sessão de exercício, a equipe envolvida no estudo dará todo o suporte necessário. Além disso, pode acontecer de você ficar cansado ou incomodado ao responder os questionários da pesquisa, mas, nestes casos, você poderá solicitar uma pausa para descansar a qualquer momento que julgar necessário. Ainda, as sessões de exercício serão conduzidas por profissionais capacitados, que te instruirão adequadamente quanto à realização de cada atividade e te darão todo o suporte necessário ao longo de todo o estudo.

**Benefícios esperados:** Como benefícios, o(a) senhor(a) receberá uma avaliação ampla da sua saúde cardiovascular, mental, cognitiva e clínica, além da prescrição e supervisão da modalidade Yoga com enfoque em melhoria dos prejuízos ocasionados pela Hipertensão Arterial.

Retirada do Consentimento: O senhor(a) pode retirar seu consentimento e desistir de participar da pesquisa a qualquer momento, sem qualquer prejuízo.

Garantia do Sigilo e de Indenização: As informações obtidas nesta pesquisa serão analisadas em conjunto com as de outros participantes, não sendo divulgado sua identificação em nenhum momento. No entanto, é importante informar que existe remota possibilidade da quebra do sigilo de maneira involuntária e não intencional (por exemplo, perda ou roubo de documentos, computadores, softwares, pendrive) e, nessa situação, as consequências serão tratadas nos termos da lei. O(a) senhor(a) poderá, quando quiser, ter acesso às informações constantes nesta declaração ou a qualquer outra informação que deseje sobre este estudo, incluindo os resultados de seus exames. Não há nenhum tipo de custos para o senhor(a) relacionado aos exames, consultas ou intervenção deste projeto. Também não há compensação financeira relacionada à sua participação. Se existir qualquer despesa adicional relacionada aos procedimentos experimentais e participação no estudo, a equipe de pesquisa fará o ressarcimento. Os dados coletados serão utilizados exclusivamente para os fins desta pesquisa. Ademais, diante de eventuais danos materiais ou imateriais provenientes da pesquisa, o(a) senhor(a) terá direito à indenização conforme preconiza a resolução vigente.

O Comitê de Ética em Pesquisa (CEP) é um colegiado interdisciplinar e independente, que deve existir nas instituições que realizam pesquisas envolvendo seres humanos no Brasil, criado para defender os interesses dos participantes de pesquisas em sua integridade e dignidade e para contribuir no desenvolvimento das pesquisas dentro dos padrões éticos (Normas e Diretrizes Regulamentadoras da Pesquisa envolvendo Seres Humanos – Res. CNS nº 466/12).

O CEP é responsável pela avaliação e acompanhamento dos protocolos de pesquisa no que corresponde aos aspectos éticos.

Endereço do CEP da Universidade Federal de Santa Catarina: Prédio Reitoria II R: Desembargador Vitor Lima, nº 222, sala 401, Trindade, Florianópolis/SC. CEP 88.040-400. Contato: (48) 3721-6094. E-mail: cep.propesq@contato.ufsc.br

Após estes esclarecimentos, solicitamos o seu consentimento para participar desta pesquisa. Duas vias deste documento foram elaboradas e serão rubricadas e assinadas pelo(a) senhor(a) e pelo pesquisador responsável, sendo que uma destas vias devidamente assinada ficará com o(a) senhor(a).

Em qualquer etapa do estudo, você terá acesso aos profissionais responsáveis pela pesquisa para esclarecimento de dúvidas.

| Assinatura do Participante | |
|----------------------------|------------------------------|
| Data:/ | |
| | _ (pesquisador responsável), |
| _ | Data:/ |

- a) A ética em pesquisa implica o respeito pela dignidade humana e a proteção devida aos participantes das pesquisas científicas envolvendo seres humanos;
- b) Este estudo tem mérito científico e a equipe de profissionais envolvidos é treinada, capacitada e competente para executar os procedimentos descritos neste termo;
- c) Esta pesquisa está pautada na Resolução 466/2012, do Conselho Nacional de Saúde e os pesquisadores comprometem-se em cumprir todos os seus itens.

Prof<sup>a</sup>. Dr<sup>a</sup>. Aline Mendes Gerage (UFSC)

Tel: (48) 3721-3860

e-mail: <u>alinegerage@yahoo.com.br</u>

Endereço: Rua Itapiranga, nº 156, apto 901C, Itacorubi, Florianópolis – SC.

# ANNEX ANNEX A – EQ5D5L



## Versão em português para o Brasil

(Portuguese version for Brazil)

## VERSÃO PARA ADMINISTRAÇÃO DO ENTREVISTADOR

Observação para o entrevistador: embora deva-se considerar o estilo particular de falar do entrevistador, o texto das instruções do questionário deve ser seguido da forma mais fiel possível. No caso do sistema descritivo EQ-5D-5L na página 2 do questionário, o texto exato deve ser seguido.

Se o entrevistado tiver dificuldade em escolher uma resposta ou pedir esclarecimento, o entrevistador deve repetir a pergunta palavra por palavra e pedir ao entrevistado que responda da maneira que mais se assemelhe à sua opinião sobre sua saúde hoje.

#### INTRODUÇÃO

(Observação para o entrevistador: leia a seguinte informação para o entrevistado.)

Estamos tentando saber o que você acha sobre sua saúde. Vou explicar o que fazer à medida que formos avançando, mas peço que me interrompa se você não entender algo ou se as coisas não estiverem claras para você. Não há respostas certas ou erradas. Estamos interessados apenas na sua visão pessoal.

Primeiro, vou ler algumas perguntas. Cada pergunta tem cinco opções de resposta. Digame qual resposta melhor descreve sua saúde HOJE.

Não escolha mais de uma resposta para cada grupo de perguntas.

(Observação para o entrevistador: leia primeiro as cinco alternativas para cada pergunta. Em seguida, peça para o entrevistado escolher qual delas se aplica a seu caso. Repita a pergunta e as alternativas, se necessário. Marque a caixa correspondente em cada cabeçalho. Talvez seja necessário lembrar o entrevistado de tempos em tempos que o período de referência é HOJE.)

#### SISTEMA DESCRITIVO EQ-5D

Primeiro, gostaria de perguntar-lhe sobre MOBILIDADE. Você diria que:

| Não tem problemas para andar? | |
|---|---|
| Tem problemas <u>leves</u> para andar? | |
| Tem problemas <u>moderados</u> para andar? | |
| Tem problemas graves para andar? | |
| É <u>incapaz</u> de andar? | |
| Agora, gostaria de perguntar-lhe sobre os CUIDADOS PESSOAIS. Você diria q | ue: |
| 1. <u>Não</u> tem problemas para se lavar ou se vestir? | |
| Tem problemas <u>leves</u> para se lavar ou se vestir? | |
| Tem problemas <u>moderados</u> para se lavar ou se vestir? | |
| Tem problemas graves para se lavar ou se vestir? | |
| É <u>incapaz</u> de se lavar ou se vestir? | |
| Agora, gostaria de perguntar-lhe sobre as ATIVIDADES HABITUAIS, como trabestudos, atividades domésticas, atividades em família ou de lazer. Você diria d | |
| 1. <u>Não</u> tem problemas para realizar as suas atividades habituais? | |
| Tem problemas <u>leves</u> para realizar as suas atividades habituais? | |
| Tem problemas moderados para realizar as suas atividades habituais? | |
| Tem problemas graves para realizar as suas atividades habituais? | |
| É <u>incapaz</u> de realizar as suas atividades habituais? | |
| Agora, gostaria de perguntar-lhe sobre DOR OU MAL-ESTAR. Você diria que: | |
| 1. Não tem dores ou mal-estar? | |
| Tem dores ou mal-estar leves? | |
| Tem dores ou mal-estar moderados? | |
| Tem dores ou mal-estar fortes? | |
| Tem dores ou mal-estar extremos? | |
| Por último, gostaria de perguntar-lhe sobre ANSIEDADE OU DEPRESSÃO. Vo | cê diria que: |
| 1. <u>Não</u> está ansioso/a ou deprimido/a? | |
| Está <u>levemente</u> ansioso/a ou deprimido/a? | |
| Está moderadamente ansioso/a ou deprimido/a? | |
| Está <u>muito</u> ansioso/a ou deprimido/a? | |
| Está extremamente ansioso/a ou deprimido/a? | |

## **EQ-5D VAS**

- Agora, eu gostaria de perguntar-lhe o quanto sua saúde está boa ou ruim HOJE.
- Gostaria que você imaginasse em sua mente uma linha vertical numerada de 0 a 100.

(Observação para o entrevistador: se estiver entrevistando pessoalmente, mostre a linha VAS para o entrevistado.)

- 100 na parte superior da linha significa a melhor saúde que você possa imaginar.
- 0 na parte inferior da linha significa a <u>pior</u> saúde que você possa imaginar.
- Agora, gostaria que você me dissesse o ponto nessa linha em que você colocaria sua saúde HOJE. (Observação para o entrevistador: marque a linha no ponto correspondente à saúde hoje do entrevistado. Agora, escreva na caixa abaixo o número que você marcou na linha.)



Obrigado por dedicar seu tempo para responder a estas perguntas.

A pior

saúde que você

### ANNEX B - SF-36

## Versão Brasileira do Questionário de Qualidade de Vida -SF-36

## 1- Em geral você diria que sua saúde é:

| Excelente | Muito Boa | Boa | Ruim | Muito Ruim |
|-----------|-----------|-----|------|------------|
| 1 | 2 | 3 | 4 | 5 |

2- Comparada há um ano atrás, como você se classificaria sua idade em geral, agora?

| Muito Melhor | Um Pouco Melhor | Quase a Mesma | Um Pouco Pior | Muito Pior |
|--------------|-----------------|---------------|---------------|------------|
| 1 | 2 | 3 | 4 | 5 |

3- Os seguintes itens são sobre atividades que você poderia fazer atualmente durante um dia comum. Devido à sua saúde, você teria dificuldade para fazer estas atividades? Neste caso, quando?

| Atividades | Sim, dificulta<br>muito | Sim, dificulta<br>um pouco | Não, não<br>dificulta de<br>modo algum |
|---|---|---|---|
| a) Atividades Rigorosas, que exigem<br>muito esforço, tais como correr,<br>levantar objetos pesados, participar em<br>esportes árduos. | 1 | 2 | 3 |
| b) Atividades moderadas, tais como mover uma mesa, passar aspirador de pó, jogar bola, varrer a casa. | 1 | 2 | 3 |
| c) Levantar ou carregar mantimentos | 1 | 2 | 3 |
| d) Subir vários lances de escada | 1 | 2 | 3 |
| e) Subir um lance de escada | 1 | 2 | 3 |
| f) Curvar-se, ajoelhar-se ou dobrar-se | 1 | 2 | 3 |
| g) Andar mais de 1 quilômetro | 1 | 2 | 3 |
| h) Andar vários quarteirões | 1 | 2 | 3 |
| i) Andar um quarteirão | 1 | 2 | 3 |
| j) Tomar banho ou vestir-se | 1 | 2 | 3 |

4- Durante as últimas 4 semanas, você teve algum dos seguintes problemas com seu trabalho ou com alguma atividade regular, como conseqüência de sua saúde física?

| | Sim | Não |
|---|---|---|
| a) Você diminui a quantidade de tempo que se dedicava ao seu | 1 | 2 |
| trabalho ou a outras atividades? | | |
| b) Realizou menos tarefas do que você gostaria? | 1 | 2 |
| c) Esteve limitado no seu tipo de trabalho ou a outras atividades. | 1 | 2 |
| d) Teve dificuldade de fazer seu trabalho ou outras atividades (p. | 1 | 2 |
| ex. necessitou de um esforço extra). | | |

5- Durante as últimas 4 semanas, você teve algum dos seguintes problemas com seu trabalho ou outra atividade regular diária, como conseqüência de algum problema emocional (como se sentir deprimido ou ansioso)?

| | Sim | Não |
|------------------------------------------------------------------|-----|-----|
| a) Você diminui a quantidade de tempo que se dedicava ao seu | 1 | 2 |
| trabalho ou a outras atividades? | | |
| b) Realizou menos tarefas do que você gostaria? | 1 | 2 |
| c) Não realizou ou fez qualquer das atividades com tanto cuidado | 1 | 2 |
| como geralmente faz. | | |

6- Durante as últimas 4 semanas, de que maneira sua saúde física ou problemas emocionais interferiram nas suas atividades sociais normais, em relação à família, amigos ou em grupo?

| De forma nenhuma | Ligeiramente | Moderadamente | Bastante | Extremamente |
|------------------|--------------|---------------|----------|--------------|
| 1 | 2 | 3 | 4 | 5 |

7- Quanta dor no corpo você teve durante as últimas 4 semanas?

| Nenhuma | Muito leve | Leve | Moderada | Grave | Muito grave |
|---------|------------|------|----------|-------|-------------|
| 1 | 2 | 3 | 4 | 5 | 6 |

8- Durante as últimas 4 semanas, quanto a dor interferiu com seu trabalho normal (incluindo o trabalho dentro de casa)?

| De maneira alguma | Um pouco | Moderadamente | Bastante | Extremamente |
|-------------------|----------|---------------|----------|--------------|
| 1 | 2 | 3 | 4 | 5 |

9- Estas questões são sobre como você se sente e como tudo tem acontecido com você durante as últimas 4 semanas. Para cada questão, por favor dê uma resposta que mais se aproxime de maneira como você se sente, em relação às últimas 4 semanas.

| | Todo<br>Tempo | A maior parte do tempo | Uma boa<br>parte do<br>tempo | Alguma parte do tempo | Uma<br>pequena<br>parte do<br>tempo | Nunca |
|---|---|---|---|---|---|---|
| a) Quanto tempo você<br>tem se sentindo cheio de<br>vigor, de vontade, de<br>força? | 1 | 2 | 3 | 4 | 5 | 6 |
| b) Quanto tempo você tem se sentido uma pessoa muito nervosa? | 1 | 2 | 3 | 4 | 5 | 6 |
| c) Quanto tempo você<br>tem se sentido tão<br>deprimido que nada<br>pode anima-lo? | 1 | 2 | 3 | 4 | 5 | 6 |
| d) Quanto tempo você tem se sentido calmo ou tranquilo? | 1 | 2 | 3 | 4 | 5 | 6 |

| e) Quanto tempo você<br>tem se sentido com<br>muita energia? | 1 | 2 | 3 | 4 | 5 | 6 |
|---|---|---|---|---|---|---|
| f) Quanto tempo você<br>tem se sentido<br>desanimado ou abatido? | 1 | 2 | 3 | 4 | 5 | 6 |
| g) Quanto tempo você<br>tem se sentido<br>esgotado? | 1 | 2 | 3 | 4 | 5 | 6 |
| h) Quanto tempo você<br>tem se sentido uma<br>pessoa feliz? | 1 | 2 | 3 | 4 | 5 | 6 |
| i) Quanto tempo você tem se sentido cansado? | 1 | 2 | 3 | 4 | 5 | 6 |

10 Durante as últimas 4 semanas, quanto de seu tempo a sua saúde física ou problemas emocionais interferiram com as suas atividades sociais (como visitar amigos, parentes, etc)?

| Todo | A maior parte do | Alguma parte do | Uma pequena | Nenhuma parte |
|-------|------------------|-----------------|----------------|---------------|
| Tempo | tempo | tempo | parte do tempo | do tempo |
| 1 | 2 | 3 | 4 | 5 |

11 O quanto verdadeiro ou falso é cada uma das afirmações para você?

| | Definitivamente verdadeiro | A maioria<br>das vezes<br>verdadeiro | Não<br>sei | A maioria<br>das vezes<br>falso | Definitiva-<br>mente falso |
|---|---|---|---|---|---|
| a) Eu costumo obedecer<br>um pouco mais<br>facilmente que as outras<br>pessoas | 1 | 2 | 3 | 4 | 5 |
| b) Eu sou tão saudável<br>quanto qualquer pessoa<br>que eu conheço | 1 | 2 | 3 | 4 | 5 |
| c) Eu acho que a minha saúde vai piorar | 1 | 2 | 3 | 4 | 5 |
| d) Minha saúde é excelente | 1 | 2 | 3 | 4 | 5 |

## ANNEX C - PSQI

# Índice de qualidade de sono de Pittsburgh (PSQI-BR)

| | s aos seus hábitos de sono durante o último mês somente. Suas respostas<br>ata da maioria dos dias e noites do último mês. Por favor, responda a todas |
|---|---|
| 1. Durante o último mês, quando vo<br>Hora usual de deitar | |
| 2. Durante o último mês, quanto ter<br>Número de minutos | mpo (em minutos) você geralmente levou para dormir? |
| 3. Durante o último mês, quando vo<br>Hora usual de levantar | |
| 4. Durante o último mês, quantas ho você ficou na cama). Horas de sono por noite | oras de sono você teve? (Este pode ser diferente do número de horas que |
| Para cada uma das questões restante | es, marque a melhor (uma) resposta. Por favor, responda a todas as questões. |
| 5. Durante o último mês, com que f você | requência você teve dificuldade de dormir porque |
| (a) Não conseguiu adormecer em | até 30 minutos |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| Nenhuma no último mês<br>1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (b) Acordou no meio da noite ou d | le manhã cedo |
| Nenhuma no último mês<br>1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (c) Precisou levantar para ir ao b | anheiro |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (d) Não conseguiu respirar confor | tavelmente |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (e) Tossiu ou roncou forte | |

Menos de 1 vez/ semana \_\_\_\_\_ 3 ou mais vezes/ semana \_\_\_\_\_

Menos de 1 vez/ semana \_\_\_\_\_

Nenhuma no último mês \_\_\_\_\_

Nenhuma no último mês \_\_\_\_\_

1 ou 2 vezes/ semana \_\_\_\_\_

(f) Sentiu muito frio

| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
|---|---|
| (g) Sentiu muito calor | |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (h) Teve sonhos ruins | |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (i) Teve dor | |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| (j) Outra(s) razão (ões), por fav | or, descreva |
| | último mês, você teve dificuldade para dormir devido |
| | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana 3 | ou mais vezes/ semana |
| maneira geral? Muito boa Boa | você classificaria a qualidade do seu sono de uma |
| Ruim<br>Muito ruim | |
| "por conta própria") para lhe a | que frequência você tomou medicamento (prescrito ou<br>njudar a dormir? Menos de 1 vez/ semana 3 ou mais vezes/ semana |
| | quência você teve dificuldade de ficar acordado icipava de uma atividade social (festa, reunião de |
| Nenhuma no último mês | Menos de 1 vez/ semana |
| 1 ou 2 vezes/ semana | 3 ou mais vezes/ semana |
| 9. Durante o último mês, quão j<br>(ânimo) para fazer as coisas (su<br>Nenhuma dificuldade<br>Um problema leve<br>Um problema razoável<br>Um grande problema | problemático foi para você manter o entusiasmo<br>nas atividades habituais)? |

## ANNEX D – PHQ9

# QUESTIONÁRIO SOBRE A SAÚDE DO/A PACIENTE-(PHQ-9)

| Durante as últimas 2 sema<br>foi incomodado/a por qual<br>abaixo?<br>(Marque sua resposta com " | ACT - ACC - | Nenhuma<br>vez | Vários<br>dias | Mais da<br>metade<br>dos dias | Quase<br>todos os<br>dias |
|---|---|---|---|---|---|
| 1. Pouco interesse ou pouco | prazer em fazer as coisas | 0 | 1 | 2 | 3 |
| 2. Se sentir "para baixo", de | primido/a ou sem perspectiva | 0 | 1 | 2 | 3 |
| Dificuldade para pegar no ou dormir mais do que de | sono ou permanecer dormindo, costume | 0 | 1 | 2 | 3 |
| 4. Se sentir cansado/a ou co | om pouca energia | 0 | 1 | 2 | 3 |
| 5. Falta de apetite ou comer | ndo demais | 0 | 1 | 2 | 3 |
| | smo/a — ou achar que você é um<br>nou sua família ou você mesmo/a | 0 | 1 | 2 | 3 |
| 7. Dificuldade para se conce<br>ou ver televisão | entrar nas coisas, como ler o jornal | 0 | 1 | 2 | 3 |
| pessoas perceberem? Ou | ntar ou falar, a ponto das outras<br>u o oposto – estar tão agitado/a ou<br>andando de um lado para o outro<br>tume | 0 | 1 | 2 | 3 |
| 9. Pensar em se ferir de alguestar morto/a | uma maneira ou que seria melhor | 0 | 1 | 2 | 3 |
| | For office co | ding <u>0</u> - | + | +<br>=Total Sco | +<br>ore: |
| Se você assinalou <u>qualque</u><br>causaram para realizar set<br>pessoas? | <u>er</u> um dos problemas, indique o<br>u trabalho, tomar conta das cois | grau de <u>difi</u><br>as em casa | culdade o<br>ou para s | que os mes<br>se relaciona | mos lhe<br>ar com as |
| Nenhuma<br>dificuldade<br>□ | Alguma<br>dificuldade dif | Muita<br>Ficuldade<br>□ | | Extre<br>dificulo | ST (1993) |

Desenvolvido pelos Drs. Robert L. Spitzer, Janet B.W. Williams, Kurt Kroenke e colegas, com um subsídio educacional da Pfizer Inc. Não é necessária permissão para reproduzir, traduzir, exibir ou distribuir.
### ANNEX E - ESCALA HOSPITAL ANXIETY AND DEPRESSION (HAD)

Este questionário ajudará o seu médico a saber como você está se sentindo. Leia todas as frases. Marque com um "X" a resposta que melhor corresponder a como você tem se sentido na última semana. Não é preciso ficar pensando muito em cada questão. Neste questionário as respostas espontâneas têm mais valor do que aquelas em que se pensa muito. Marque apenas uma resposta para cada pergunta.

| 1A. Eu me sinto tenso ou contraído:<br>( 3 ) A maior parte do tempo<br>( 2 ) Boa parte do tempo | (1)De vez em quando<br>(0)Nunca |
|---|---|
| 2D. Eu ainda sinto gosto pelas mesmas coisas de antes:<br>( 0 ) Sim, do mesmo jeito que antes<br>( 1 ) Não tanto quanto antes | (2)Só um pouco<br>(3)Já não sinto mais prazer em nada |
| 3A. Eu sinto uma espécie de medo, como se alguma coisa ruim<br>( 3 ) Sim, e de um jeito muito forte<br>( 2 ) Sim, mas não tão forte | fosse acontecer: ( 1 ) Um pouco, mas isso não me preocupa ( 0 ) Não sinto nada disso |
| 4D. Dou risada e me divirto quando vejo coisas engraçadas:<br>( 0 ) Do mesmo jeito que antes<br>( 1 ) Atualmente um pouco menos | ( 2 ) Atualmente bem menos<br>( 3 ) Não consigo mais |
| 5A. Estou com a cabeça cheia de preocupações:<br>( 3 ) A maior parte do tempo<br>( 2 ) Boa parte do tempo | (1)De vez em quando<br>(0)Raramente |
| 6D. Eu me sinto alegre:<br>( 3 ) Nunca<br>( 2 ) Poucas vezes | ( 1 ) Muitas vezes<br>( 0 ) A maior parte do tempo |
| 7A. Consigo ficar sentado à vontade e me sentir relaxado:<br>( 0 ) Sim, quase sempre<br>( 1 ) Muitas vezes | ( 2 ) Poucas vezes<br>( 3 ) Nunca |
| 8D. Eu estou lento para pensar e fazer as coisas<br>( 3 ) Quase sempre<br>( 2 ) Muitas vezes | (1)De vez em quando<br>(0)Nunca |
| 9A. Eu tenho uma sensação ruim de medo, como um frio na bar<br>( 0 ) Nunca<br>( 1 ) De vez em quando | riga ou um aperto no estômago:<br>(2)Muitas vezes<br>(3)Quase sempre |
| 10D. Eu perdi o interesse em cuidar da minha aparência:<br>( 3 ) Completamente<br>( 2 ) Não estou mais me cuidando como eu deveria | ( 1 ) Talvez não tanto quanto antes<br>( 0 ) Me cuido do mesmo jeito que antes |
| 11A. Eu me sinto inquieto, como se eu não pudesse ficar parado<br>( 3 ) Sim, demais<br>( 2 ) Bastante | o em lugar nenhum:<br>(1)Um pouco<br>(0)Não me sinto assim |
| 12D. Fico esperando animado as coisas boas que estão por vir ( 0 ) Do mesmo jeito que antes ( 1 ) Um pouco menos do que antes | ( 2 ) Bem menos do que antes<br>( 3 ) Quase nunca |
| 13A. De repente, tenho a sensação de entrar em pânico: | |

| ( 3 ) A quase todo o momento<br>( 2 ) Várias vezes | ( 1 ) De vez em quando<br>( 0 ) Não sinto isso |
|---|---|
| 14D. Consigo sentir prazer quando assisto um bom programa d | e televisão, de rádio, ou quando leio alguma coisa: |
| ( 0 ) Quase sempre<br>( 1 ) Várias vezes<br>( 2 ) Pouca vezes<br>( 3 ) Quase nunca | |

#### ANNEX F - PSS-10

## ESCALA DE PERCEPÇÃO DE ESTRESSE-10 (EPS-10)

As questões nesta escala perguntam a respeito dos seus sentimentos e pensamentos durantes os últimos 30 dias (último mês). Em cada questão indique a freqüência com que você se sentiu ou pensou a respeito da situação.

| | | 40.0 | о произона на | | |
|---|---|---|---|---|---|
| 1. | | eqüência você fi<br>esperadamente? (c | | do por causa de<br>imos 30 dias) | algo que |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 2. | | üência você senti<br>a sua vida? (consi | | apaz de controlar<br>s 30 dias) | coisas |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 3. | Com que frequé dias) | ência você esteve n | ervoso ou estre | essado? (considere c | s últimos 30 |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 4. | • | qüência você este<br>oblemas pessoais? ( | | em sua capacidad<br>Iltimos 30 dias) | e de lidar |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 5. | | üência você se<br>erava? (considere | • | oisas aconteceram d<br>dias) | la maneira |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 6. | | ência você achou d<br>fazer? (considere d | • | guiria lidar com toda<br>ias) | s as coisas |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [4] Muito |
| 7. | • | μüência você foi α<br>últimos 30 dias) | capaz de cont | trolar irritações na | sua vida? |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 8. | | iência você sentiu<br>(considere os últin | | aspectos de sua vic | la estavam |
| | [ 0 ].Nunca<br>Freqüente | [ 1 ].Quase Nunca | [ 2 ].Às Vezes | [ 3 ].Pouco Freqüente | [ 4 ] Muito |
| 9. | | üência você estev<br>ontrole? (considere | • | ausa de coisas que<br>dias) | estiveram |

10. Com que freqüência você sentiu que os problemas acumularam tanto que você não conseguiria resolvê-los? (considere os últimos 30 dias)

#### ANNEX G - MoCa

"Este é um teste para avaliar suas capacidades cognitivas. Fique tranquilo e seja preciso em suas respostas".

#### 1. Alternância de trilha

<u>Aplicação</u>: "Desenhe uma linha indo de um número para uma letra em ordem crescente. Comece aqui {aponte para (1)} e desenhe uma linha de 1 para A, daí para 2 e assim por diante. Termine aqui {aponte para (E)}."

Pontuação: 1 ponto se o sujeito desenhar o padrão, sem desenhar nenhuma linha que ultrapasse o alvo.

#### 2. Habilidades Viso-Construtivas (Cubo)

Aplicação: (Apontando para o cubo) "Copie este desenho o mais precisamente que você puder, no espaço abaixo" Pontuação: 1 ponto para a execução correta do desenho (tridimensional, sem adição ou ausência de linha ou linhas de comprimento diferente).

#### 3. Habilidades Viso-Construtivas (Relógio)

Aplicação: (Indique o espaço) "Desenhe um relógio. Coloque todos os números e marque a hora 11:10"

Pontuação: Contorno, Números e Ponteiros (1 ponto)

#### 4. Nomeação

Aplicação: Começando à esquerda, aponte para cada figura e diga: "Me diga o nome desse animal" Pontuação: Cada ponto é dado para as respostas: (1) rinoceronte, (2) leão, (3) camelo ou dromedário

#### 5. Memória

Aplicação: "Este é um teste de memória. Eu lerei uma lista de palavras que você deverá lembrar-se agora e mais tarde. Ouça com muita atenção. Quando eu terminar, me diga todas as palavras que você lembrar."

Quando o sujeito indicar que terminou (lembrou-se de todas as palavras), ou que não se lembra de mais nenhuma palavra, leia a lista pela segunda vez com as seguintes instruções: "Eu lerei a mesma lista pela segunda vez. Tente se lembrar e me diga todas as palavras que você puder, incluindo palavras ditas da primeira vez." final da segunda tentativa, informe o sujeito que lhe será pedido para resgatar essas palavras novamente, dizendo: "Memorize estas palavras pois eu lhe pedirei para resgatar essas palavras novamente no final do teste."

Pontuação: Não são dados pontos neste momento, a memória é avaliada lá no final do teste

#### 6. Atenção

#### Span de dígitos direto

<u>Aplicação</u>: "Eu lhe direi alguns números e quando eu terminar, me repita na mesma ordem exata que eu disse." Leia a sequência de 5 números no intervalo de um dígito por segundo.

Pontuação: Atribua um ponto para cada seqüência repetida corretamente.

#### Span de dígitos indireto

Aplicação: "Agora eu vou ler mais alguns números porém, você vai repeti-los na ordem inversa."

Pontuação: Atribua um ponto para cada sequência repetida corretamente.

#### Vigilância

Aplicação: "Agora vou ler uma seqüência de letras. Toda a vez que eu disser a letra A, bata a mão na mesa. Se eu disser uma letra diferente, não bata a sua mão."

Pontuação: Dê 1 ponto de zero a um erro e 0 pontos se houver 2 ou mais erros

#### **Sete Seriado**

Aplicação: "Agora eu lhe pedirei para que você subtraia sete a partir de 100, e então siga subtraindo sete da sua resposta até eu lhe disser que pare." Dê esta instrução 2 vezes se necessário. OBS: Se o voluntário errar um dos números, repita o número correto que seria correto da seguinte maneira: 93 menos 7 ou 86 menos 7.

Pontuação: Este item é pontuado com 3 pontos.

#### 7. Replicação de sentença

Aplicação: "Eu vou ler uma sentença para você. Repita depois de mim, exatamente como eu disser: Eu somente sei que João é quem será ajudado hoje." Após a resposta, diga: "Agora eu vou ler outra sentença. Repita-a depois de mim, exatamente como eu disser [pausa]: o gato sempre se esconde debaixo do sofá quando o cachorro está na sala."

Pontuação: Atribua 1 ponto para cada sentença repetida exatamente como foi lida. Esteja atento para erros que são omissões (omitir "somente", "sempre") e substituições/adições ("João é quem ajudou hoje)

#### 8. Fluência Verbal

Aplicação: "Diga-me em um minuto todas as palavras com uma certa letra do alfabeto. Você pode dizer qualquer tipo de palavra, exceto nomes próprios (como Beto ou Bráulio), números, ou palavras que começam com sons iguais porém com diferente sufixo, por exemplo, amor, amante, amando". Eu direi para parar após 1 minuto. Você está pronto? Agora, me diga quantas palavras você pode pensar que começam com a letra F". Após 1 minuto, interrompa. Pontuação: Atribua 1 ponto se o sujeito gerar 11 palavras ou mais em 60 segundos. Grave a resposta do sujeito no espaço ou ao lado.

#### 9. Abstração

<u>Aplicação</u>: "Diga-me em que uma laranja e uma banana são parecidas". Se o sujeito responde de maneira errada, diga somente uma vez adicional: "Me diga de outra forma em que estes 2 itens são parecidos". Se o sujeito não der a resposta apropriada (fruta), diga, "sim, e elas são ambas frutas" não dê nenhuma outra instrução ou esclarecimento.

Após o ensaio, diga: "Agora me diga em que um trem e uma bicicleta são parecidos". Após a resposta, aplique a segunda tentativa dizendo: "Agora me diga em que uma régua e um relógio são parecidos". Não dê nenhuma instrução adicional ou dica.

<u>Pontuação</u>: Dê 1 ponto para cada par de itens corretamente respondidos (banana e laranja não são pontuados). As seguintes respostas são aceitas; trem-bicicleta=meios de transporte, meios de viajar, você viaja em ambos; réguarelógio=instrumentos de medida, usados para medir. As seguintes respostas não são aceitas: trem-bicicleta=eles têm rodas; régua-relógio=eles têm números.

#### 10. Evocação Tardia

Aplicação: "Se lembra que anteriormente eu li algumas palavras para você, as quais eu pedi que você se lembrasse. Me diga quantas dessas palavras você pode lembrar." Faça uma marca  $(\sqrt{})$  para cada uma das palavras lembradas corretamente espontaneamente sem nenhuma pista, no espaço alocado.

Pontuação: Atribua 1 ponto para cada palavra lembrada livremente sem nenhuma pista.

#### 11. Orientação

Aplicação: "Diga-me a data de hoje". Se o sujeito não der a resposta correta, então diga imediatamente:" Me diga [o ano, mês, data exata e o dia da semana]". Então diga: "Agora me diga o nome deste lugar e em que cidade fica". Pontuação: Atribua 1 ponto para cada item corretamente respondido. O sujeito deve dizer a data e local exatos (nome do hospital, setor, consultório). Não são atribuídos pontos se o sujeito comete erro de um dia para outro dia e a data.

**Resultado Total**: Some todos os resultados listados à margem direita. Adicione 1 ponto para o indivíduo que possui 12 anos de escolaridade formal (caso tenha até o "científico" ou "ensino médio completo").

#### ANNEX H – Stroop Color Test

"Agora faremos um teste de atenção. Nesta tarefa as palavras (verde, vermelho, azul e amarelo) estão escritas em cores distintas (verde, vermelho, azul e amarelo) como se vê no modelo adaptado abaixo".

•

#### I) Primeiramente você será instruído a falar a palavra que está escrita:

Mostre a primeira linha da folha de respostas e confira as respostas abaixo:

| VERDE VERMELHO | AZUL | VERMELHO | AZUL |
|----------------|------|----------|------|
|----------------|------|----------|------|

#### II) Agora, você irá me falar de que cor que está escrito:

Mostre a primeira linha da folha de respostas e confira as respostas abaixo:

| AMARELO VERMELHO | VERMELHO | AMARELO | VERMELHO |
|------------------|----------|---------|----------|
|------------------|----------|---------|----------|

<sup>\*</sup>Em caso de erros durante a prévia o aplicador deve imediatamente fornecer a resposta correta.

"Terminado esse teste, agora você deverá me dizer a cor escrita de todas as 40 palavras contidas na folha no menor tempo possível e com a menor quantidade de erros (os quais serão corrigidos)"

Na segunda parte (incongruente), você deverá me dizer a cor que cada das 40 palavras contidas na folha está escrita. Isso deve ser feito no menor tempo possível e com a menor quantidade de erros (os quais serão corrigidos).

Caso o avaliado acerte o primeiro número da sequência de 2 à 9 números, pular para a sequência com .Caso o voluntário erre as duas tentativas do 'span' o teste é finalizado e o 'span máximo' será referente à classe anterior. Em outras palavras, no primeiro erro cometido em determinado 'span' é lida a outra sequência da classe, e caso o sujeito acerte é repetida a sequência na qual foi cometido o erro. Acertando irá para a próxima classe, errando o teste se encerra).

<sup>\*</sup>Cada erro durante a fase de testagem deve ser imediatamente sinalizado pelo aplicador e solicitada a correção além de ser registrado no quadro de respostas (como: E).

<sup>\*</sup>Deve-se cronometrar e registrado o tempo total dispendido para a execução da tarefa, o número de palavras respondidas e também o número de erros.

<sup>\*</sup>Fazer cada tomada de palavras em cada uma das partes após fazer o teste anterior logo abaixo.

# ANNEX I – Escala de Adesão Terapêutica de Morisky

# ESCALA DE ADESÃO TERAPÊUTICA DE MORISKY DE 8 ITENS (MMAS-8).

| Nome | |
|---|---|
| completo: | ID: |
| <br>Data: | Horário: |
| Avaliador: | |
| 1) Você às vezes esquece | de tomar os seus remédios para pressão? |
| ( ) Sim ( ) Não | |
| 2) Nas duas últimas semar | nas, houve algum dia em que você não tomou seus |
| remédios para pressão alta? | |
| ( ) Sim ( ) Não | |
| 3) Você já parou de tomar se | eus remédios ou diminuiu a dose sem avisar seu médico |
| porque se sentia pior quando o | os tomava? |
| ( ) Sim ( ) Não | |
| 4) Quando você viaja ou sai | de casa, às vezes esquece de levar seus medicamentos? |
| ( ) Sim ( ) Não | |
| 5) Você tomou seus medicar | mentos para pressão alta ontem? |
| ( ) Sim ( ) Não | |
| 6) Quando sente que sua pre | essão está controlada, você às vezes para de tomar seus |
| medicamentos? | |
| ( ) Sim ( ) Não | |
| 7) Você já se sentiu income | odado por seguir corretamente o seu tratamento para |
| pressão alta? | |
| ( ) Sim ( ) Não | |

| 8) | Com | que frequé | ência v | ocê tem dificı | uldades | para se lembr | ar de to | omar todos os seus |
|---|---|---|---|---|---|---|---|---|
| remé | édios p | oara press | são? | | | | | |
| | ( | ) Nunca | ( | ) Quase | ( | ) Às vezes | ( | ) |
| Freq | luente | mente | ( | ) Sempre | | | | |

## ANNEX J – Questionário de Frequência Alimentar

### QUESTIONÁRIO DE FREQUÊNCIA ALIMENTAR

## QUESTIONÁRIO DE FREQUÊNCIA ALIMENTAR

Nos últimos 3 meses, com que frequência você comeu/bebeu?

| Alimento/grupo | Vezes e frequência |
|---|---|
| 1) Leite | 1.1) ( )Número vezes (88)Não se Aplica |
| | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 2) Derivados de leite (queijo, iogurte, etc.) | 2.1) ( )Número vezes (88)Não se Aplica |
| | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 3) Frutas (banana, maçã, laranja, etc.) | 3.1) ( )Número vezes (88)Não se Aplica |
| | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 4) Verduras e legumes crus ou cozidos | 4.1) ( )Número vezes (88)Não se Aplica |
| (alface, couve, cenoura, abobrinha, | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| repolho, etc.) | |
| 5) Leguminosas (feijão, lentilha, grão de | 5.1) ( )Número vezes (88)Não se Aplica |
| bico, ervilha) | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 6) Carnes em geral (boi, porco e frango) | 6.1) ( )Número vezes (88)Não se Aplica |
| | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 7) Peixe | 7.1) ( )Número vezes (88)Não se Aplica |
| 2) 2 | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 8) Ovos | 8.1) ( ) Número vezes (88) Não se Aplica |
| 0) 5 1 111 1 1 1 1 | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 9) Embutidos (salsicha, salame, linguiça, | 9.1) ( )Número vezes (88)Não se Aplica |
| presunto, etc.) | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 10) Pão, biscoitos salgados e doces | 10.1) ( )Número vezes (88)Não se Aplica |
| 11) Biscoitos recheados | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca<br>11.1) ( )Número vezes (88)Não se Aplica |
| li) biscoitos recileados | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 12) Doce, bala, chiclete e chocolate | 12.1) ( )Número vezes (88)Não se Aplica |
| 12) boce, bala, chiclete e chocolate | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 13) Salgados (coxinha,etc.), sanduíche, | 13.1) ( )Número vezes (88)Não se Aplica |
| (cachorro quente, etc.) ou salgadinhos | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| "chips" | (1)Dia (2)Schiana (S)Mics (4)Maro (S)Marica |
| 14) Refrigerantes | 14.1) ( )Número vezes (88)Não se Aplica |
| | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| | (-), (-), (-), (-), |
| 15) Tubérculos e raízes (batata, mandioca, | 15.1) ( )Número vezes (88)Não se Aplica |
| inhame, etc.) | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |
| 16) Temperos industrializados (como caldo | 16.1) ( )Número vezes (88)Não se Aplica |
| Knor, sazon) | (1)Dia (2)Semana (3)Mês (4)Raro (5)Nunca |

**ANNEX K** – Escala de Percepção de Esforço (BORG)

| Classificação | Descritor |
|---------------|--------------------|
| 0 | Repouso |
| 1 | Muito, Muito Fácil |
| 2 | Fácil |
| 3 | Moderado |
| 4 | Um Pouco Difícil |
| 5 | Difícil |
| 6 | *** |
| 7 | Muito Difícil |
| 8 | * |
| 9 | 8 |
| 10 | Máximo |

Escala CR10 de Borg (1982) modificada por Foster et. al. (2001).

**ANNEX** L – Escala de Sensação

| +5 | Muito bom |
|----|--------------------|
| +4 | |
| +3 | Razoavelmente bom |
| +2 | |
| +1 | Bom |
| 0 | Neutro |
| -1 | Ruim |
| -2 | |
| -3 | Razoavelmente ruim |
| -4 | |
| -5 | Muito ruim |

Escala de Sensação de Hardy e Rejeski (HARDY; REJESKI, 1989).